CLINICAL TRIAL: NCT00989079
Title: A Phase 1 Placebo-Controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of PF-04971729 After Administration of Single Escalating Oral Doses Under Fed and Fasted Conditions in Healthy Volunteers
Brief Title: A Single Escalating Dose Study Of Ertugliflozin (PF-04971729, MK-8835) Under Fed and Fasted Conditons In Healthy Volunteers (MK-8835-036)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 8835-036
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Single Ascending Dose Study in healthy subjects
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 Sequence 1 (Experimental): Period 1 (fasted) Placebo → Period 2 (fasted) ertugliflozin (E) 10 mg → Period 3 (fasted) E 100 mg → Period 4 (fed) E 100 mg. Each dose of study drug will be separated by a minimum of 7 days.
  Interventions: Drug: Ertugliflozin; Drug: Placebo to Ertugliflozin
- Cohort 1 Sequence 2 (Experimental): Period 1 (fasted) E 0.5 mg → Period 2 (fasted) Placebo → Period 3 (fasted) E 100 mg → Period 4 (fed) E 100 mg. Each dose of study drug will be separated by a minimum of 7 days.
  Interventions: Drug: Ertugliflozin; Drug: Placebo to Ertugliflozin
- Cohort 1 Sequence 3 (Experimental): Period 1 (fasted) E 0.5 mg → Period 2 (fasted) E 10 mg → Period 3 (fasted) Placebo → Period 4 (fed) E 100 mg. Each dose of study drug will be separated by a minimum of 7 days.
  Interventions: Drug: Ertugliflozin; Drug: Placebo to Ertugliflozin
- Cohort 2 Sequence 1 (Experimental): Period 1 (fasted) Placebo → Period 2 (fasted) E 30 mg → Period 3 (fasted) E 300 mg. Each dose of study drug will be separated by a minimum of 7 days.
  Interventions: Drug: Ertugliflozin; Drug: Placebo to Ertugliflozin
- Cohort 2 Sequence 2 (Experimental): Period 1 (fasted) E 2.5 mg → Period 2 (fasted) Placebo → Period 3 (fasted) E 300 mg. Each dose of study drug will be separated by a minimum of 7 days.
  Interventions: Drug: Ertugliflozin; Drug: Placebo to Ertugliflozin
- Cohort 2 Sequence 3 (Experimental): Period 1 (fasted) E 2.5 mg → Period 2 (fasted) E 30 mg → Period 3 (fasted) Placebo. Each dose of study drug will be separated by a minimum of 7 days.
  Interventions: Drug: Ertugliflozin; Drug: Placebo to Ertugliflozin

INTERVENTIONS:
Drug: Ertugliflozin — Ertugliflozin will be administered as an extemporaneously prepared suspension/solution for all doses within the initially planned range.
Drug: Placebo to Ertugliflozin — Correspondingly placebo doses to ertugliflozin will be administered as suspension/solution

SUMMARY:
Ertugliflozin (PF-04971729, MK-8835) is a new compound proposed for the treatment of Type 2 diabetes mellitus. The primary purpose of this study is to evaluate the safety and tolerability along with the pharmacokinetics of single escalating doses of ertugliflozin under fed and fasted conditions in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-10-16 (Actual); Primary Completion 2009-12-11 (Actual); Study Completion 2009-12-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing an Adverse Event (AE) | Up to Day 10 of each dosing period
Number of Participants Discontinuing Study Drug Due to an AE | Up to Day 8 of each dosing period
Change from baseline in 24-hour urinary glucose excretion | Baseline and 24 hours
Area under the plasma concentration-time curve (AUC) from Time 0 to infinity (AUCinf) for ertugliflozin | Up to Day 4 of each treatment period
Area under the plasma concentration-time curve (AUC) from Time 0 to time of the last quantifiable concentration (AUClast) for ertugliflozin | Up to Day 4 of each treatment period
Maximum plasma concentration (Cmax) of ertugliflozin | Up to Day 4 of each treatment period
Time taken to reach the maximum observed plasma concentration (Tmax) of ertugliflozin | Up to Day 4 of each treatment period
Ertugliflozin half life (t1/2) | Up to Day 4 of each treatment period
Apparent clearance (CL/F) after a single dose of ertugliflozin | Up to Day 4 of each treatment period
Apparent volume of distribution (Vz/F) | Up to Day 4 of each treatment period

SECONDARY OUTCOMES:
Urinary glucose excretion over 72 hours | Up to 72 hours of each dosing period
Change from baseline in 24-hour weighted mean glucose | Baseline and 24 hours
Inhibition of glucose reabsorption | Up to 24 hours of each dosing period
Renal clearance (CLr) of Ertugliflozin | Up to 24 hours of each dosing period
Urinary recovery of Ertugliflozin | Up to 24 hours of each dosing period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Fediuk DJ, Nucci G, Dawra VK, Cutler DL, Amin NB, Terra SG, Boyd RA, Krishna R, Sahasrabudhe V. Overview of the Clinical Pharmacology of Ertugliflozin, a Novel Sodium-Glucose Cotransporter 2 (SGLT2) Inhibitor. Clin Pharmacokinet. 2020 Aug;59(8):949-965. doi: 10.1007/s40262-020-00875-1. PMID 32337660
- [Derived] Fediuk DJ, Sahasrabudhe V, Dawra VK, Zhou S, Sweeney K. Population Pharmacokinetic Analyses of Ertugliflozin in Select Ethnic Populations. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1297-1306. doi: 10.1002/cpdd.970. Epub 2021 Jul 2. PMID 34213819
- [Derived] Marshall JC, Liang Y, Sahasrabudhe V, Tensfeldt T, Fediuk DJ, Zhou S, Krishna R, Dawra VK, Wood LS, Sweeney K. Meta-Analysis of Noncompartmental Pharmacokinetic Parameters of Ertugliflozin to Evaluate Dose Proportionality and UGT1A9 Polymorphism Effect on Exposure. J Clin Pharmacol. 2021 Sep;61(9):1220-1231. doi: 10.1002/jcph.1866. Epub 2021 Jun 19. PMID 33813736
- [Derived] Callegari E, Lin J, Tse S, Goosen TC, Sahasrabudhe V. Physiologically-Based Pharmacokinetic Modeling of the Drug-Drug Interaction of the UGT Substrate Ertugliflozin Following Co-Administration with the UGT Inhibitor Mefenamic Acid. CPT Pharmacometrics Syst Pharmacol. 2021 Feb;10(2):127-136. doi: 10.1002/psp4.12581. Epub 2020 Dec 30. PMID 33314761